CLINICAL TRIAL: NCT00408798
Title: Treatment of Alopecia Areata of the Scalp With Intradermal Injections of Botulinum Toxin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: H06-00278; Health Canada: Control #108512
Record Dates: First submitted 2006-12-05; First posted 2006-12-07 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-03

CONDITIONS: Alopecia Areata
Keywords: Treatment of Alopecia areata with intracutaneous injections of Botulinum Toxin A
MeSH Terms: conditions — Alopecia Areata | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Intracutaneous injections of Botulinum Toxin A (Botox), 0.1 cc per injection site, which equals 10 units — See Detailed Description.

SUMMARY:
The purpose of this study is to examine prospectively the safety and efficacy of Botulinum Toxin A (Botox) injections in the treatment of patients with alopecia areata of the scalp.

DETAILED DESCRIPTION:
Hypothesis Intralesional injections of Botulinum Toxin A can be used as a treatment for AA. Potential points of action of this treatment include changes in neurotransmitters, which either directly or via neuroimmunologic mechanisms influence cytocines that are responsible for the hair growth arrest in alopecia areata.

Justification Botulinum Toxin A is an antagonist of Acetylcholine esterase and is used to treat facial wrinkles and hyperhidrosis. One ampoule contains Clostridium Botulinum Toxin Typ A (900kD) 100 E, other components are human albumin and sodium choride. The investigator has learnt about the potential effect of this treatment in AA from personal communication.

Objectives Over a period of 6 month, to assess the therapeutic efficacy and safety of a regimen of two interlesional injections of Botulinum Toxin A at 0 and 3 months, in patients with alopecia areata of the scalp, compared to placebo.

Research Method A total of 20 eligible patients will be enrolled in the study. All patients will receive treatment into one half of their target area and placebo treatment into the other half of their target area.

Measurement of the severity of scalp alopecia areata will be based on the extent terminal scalp hair loss. The Severity of Alopecia Tool (SALT) will be used, which determines the percent of scalp involvement with disease as calculated according to specifications detailed in the Alopecia Areata Investigational Guidelines by Olsen et al..

A circular target area of at least 4 cm diameter will be chosen on the scalp.

At visit 0 and after 3 months at visit 1, the two right quandrants of the target area will each be injected with either Botulinum Toxin A (Botox) at a dose of 10 Units (0.1 cc) or saline 0.9% with a total of 0.1 cc.

The left two quadrants will be injected with the other medication. The patient will not know which half of the target area is injected with the drug or placebo.

The chosen side will be noted in the patient documentation by one investigator. The second investigator who does the efficacy assessment with the qualitative scale will not know which side is treated with Botulinum Toxin A or placebo.

At every visit, extent of the hair loss in the test area will be examined, based on a semi quantitative assessment scale ranging from 0 to 100. The investigator does not know which side had been treated.

There had been unpublished anecdotal reports of the use and the efficacy of Botulinumtoxin A in patients with alopecia areata. No further evidence is available so fare.

ELIGIBILITY:
Inclusion Criteria:

* Patients with long standing alopecia areata, patches must be at least 4 cm in diameter

Exclusion Criteria:

* Intake of drugs that interfere with Botulinum toxin A such as gentamicin, tobramycin, clindamycin and lincomycin; medications used to treat heart rhythm problems, such as quinidine; and medications used to treat other conditions, such as myasthenia gravis, ALS or Alzheimer's disease.
* Neuromuscular disorders such as Myasthenia gravis and Lambert-Eaton-Syndrome.
* Treatment with another investigational drug within 4 weeks prior to anticipated first treatment.
* Females who are pregnant, planning to become pregnant during the study period, or breastfeeding.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2007-10; Primary Completion 2009-10-30 (Actual); Study Completion 2009-10-30 (Actual)

PRIMARY OUTCOMES:
To evaluate hair regrowth with alopecia areata subcutaneous injections of Botulinum toxin A

SECONDARY OUTCOMES:
Hair regrowth will be assessed after 3 months and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jerry Shapiro, MD, FRCPC, Principal Investigator — University of British Columbia
Locations (1):
- Department of Dermatology, The Skin Care Centre, Vancouver, British Columbia, Canada